CLINICAL TRIAL: NCT02502227
Title: Mechanisms of Mindfulness Training and Stress Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Pittsburgh (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R21AT008493-01A1 (NIH)
Record Dates: First submitted 2015-07-07; First posted 2015-07-20 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Psychological Stress; Mindfulness
Keywords: mindfulness; psychological stress; wellness programs; cortisol
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mindfulness Training (Active Comparator): Mindfulness training intervention consisting of eight weekly 2.5 hour group sessions, a day-long retreat in the sixth week, and daily home mindfulness meditation
  Interventions: Behavioral: Mindfulness
- Mindful Attention Only Training (Active Comparator): Mindful attention only training intervention consisting of eight weekly 2.5 hour group sessions, a day-long retreat in the sixth week, and daily home mindfulness meditation
  Interventions: Behavioral: Mindfulness
- No Treatment Control Condition (No Intervention): No treatment participants will be informed that their participation is important and that they are requested to not seek out similar treatments during this waiting period.

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness training practices aim to foster attention and acceptance toward one's present moment experience. Mindfulness consists of two components-- (1) deploying attention to monitor one's moment-to-moment experience, and (2) fostering an attitude of acceptance toward one's moment-to-moment experience
  Arms: Mindful Attention Only Training; Mindfulness Training

SUMMARY:
This study is a three-arm randomized controlled trial of a mindfulness stress reduction intervention, with the aim of dismantling the experience-monitoring and nonjudgmental-acceptance elements of mindfulness programs to determine the active treatment component. In addition to enhancing understanding of mechanisms underlying the effects of mindfulness interventions, identifying the therapeutic constituent(s) could inform development of targeted interventions as well as provide strategies to optimize adherence.

DETAILED DESCRIPTION:
There is a growing body of randomized controlled trial (RCT) evidence indicating that mindfulness training interventions may reduce stress and improve stress-related disease outcomes. Yet little is known about the underlying active training mechanisms of mindfulness training. Although it is generally believed that mindfulness training interventions foster a capacity to monitor and accept present moment experience, debate currently focuses on whether it is the capacity to both monitor and non-judgmentally accept experience that drives the salutary effects observed in mindfulness training interventions. This project will test these putative active mechanisms by comparing two different types of mindfulness meditation training programs. N=135 stressed community adults will be recruited and randomized to either two different types of 8-week Mindfulness-Based Stress Reduction (MBSR) programs or a No Treatment Control (assessment only) comparison condition. Participants will complete 3 days of daily experience sampling (Ecological Momentary Assessment) immediately before and after the 8-week intervention period to measure attentional control and stress perceptions in daily life. In order to measure psychological and HPA-axis stress reactivity to a controlled stressor, participants will also complete a standardized acute stress challenge task (the Trier Social Stress Test, TSST) immediately following the 3-day post-intervention assessment period. This project provides the first dismantling study of mindfulness meditation training, it utilizes cutting-edge daily experience sampling of real life stress (using EMA) and stress biomarkers (salivary cortisol), and will provide important initial information for designing more effective (and efficient) mindfulness training interventions in at-risk stressed patient populations.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Moderate- to high-stress
* Owns an internet-enabled smart phone

Exclusion Criteria:

* Diagnosis of chronic mental (e.g. recurrent depression, schizophrenia, personality disorder) or physical disease (e.g. cancer, HIV, diabetes)
* Hospitalization in past 3 months
* Medication use that interferes with cortisol activity (e.g. corticosteroids)
* Current oral contraceptive use
* Pregnancy
* Current antibiotic, antiviral, or antimicrobial treatment
* Travel outside the country within the past 6 months to any country on the Center for Disease Control travel alert list
* Recreational drug use, excessive alcohol or tobacco use
* Significant experience with or daily practice of mindfulness meditation or related mind-body practice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Daily life stress assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 12 weeks

SECONDARY OUTCOMES:
Daily life state attention and acceptance assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 12 weeks
Subjective stress in response to social evaluative threat | assessed at post-intervention, which is an average of 14 weeks
Salivary Cortisol in response to social evaluative threat | assessed at post-intervention, which is an average of 14, at time 0, and 25, 35, and 60 minutes post-stress challenge
Blood Pressure reactivity to social evaluative threat (systolic and diastolic blood pressure) | assessed at post-intervention, which is an average of 14 weeks, at 2-minute intervals during session
Sustained attention measured by the Dichotic Listening Task | change from baseline to post-intervention, which is an average of 14 weeks
Sustained inattentional blindness measured by the Inattentional Blindness Task | post-intervention only

OTHER OUTCOMES:
Daily life affect assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 12 weeks
Daily life social interactions assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 12 weeks
Perceived stress using the Perceived Stress Scale | change from baseline to post-intervention, which is an average of 14 weeks
Attentional control using the Attentional Control Scale | change from baseline to post-intervention, which is an average of 14 weeks
Treatment expectancies | post-intervention an average of 14 weeks after the baseline
Subjective responses to the training program intervention | composite of ratings made after each intervention lesson, an average of 10 weeks following baseline
Mindfulness using the Mindful Attention Awareness Scale | change from baseline to post-intervention, which is an average of 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Weber, Ph.D., Study Chair — National Center for Complementary and Integrative Health, National Institutes of Health
Locations (3):
- United States (3):
  - Carnegie Mellon University, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center- Center for Integrative Medicine, Pittsburgh, Pennsylvania
  - Pennsylvania State University, University Park, Pennsylvania

REFERENCES:
- [Derived] Woods WC, Edershile EA, Ringwald WR, Sharpe BM, Himmelstein PH, Newman MG, Wilson SJ, Ellison WD, Levy KN, Pincus AL, Creswell JD, Wright AGC. Psychometric evaluation of a Visual Interpersonal Analog Scale. Psychol Assess. 2023 Apr;35(4):311-324. doi: 10.1037/pas0001210. Epub 2023 Jan 19. PMID 36656726
- [Derived] Chin B, Lindsay EK, Greco CM, Brown KW, Smyth JM, Wright AGC, Creswell JD. Mindfulness interventions improve momentary and trait measures of attentional control: Evidence from a randomized controlled trial. J Exp Psychol Gen. 2021 Apr;150(4):686-699. doi: 10.1037/xge0000969. Epub 2020 Sep 24. PMID 32969686
- [Derived] Chin B, Lindsay EK, Greco CM, Brown KW, Smyth JM, Wright AGC, Creswell JD. Psychological mechanisms driving stress resilience in mindfulness training: A randomized controlled trial. Health Psychol. 2019 Aug;38(8):759-768. doi: 10.1037/hea0000763. Epub 2019 May 23. PMID 31120272
- [Derived] Lindsay EK, Chin B, Greco CM, Young S, Brown KW, Wright AGC, Smyth JM, Burkett D, Creswell JD. How mindfulness training promotes positive emotions: Dismantling acceptance skills training in two randomized controlled trials. J Pers Soc Psychol. 2018 Dec;115(6):944-973. doi: 10.1037/pspa0000134. PMID 30550321